CLINICAL TRIAL: NCT06917755
Title: The Impact of Immersive Virtual Reality Training in Thyroid Surgery: A Prospective Randomized Controlled Trial
Brief Title: The Impact of Immersive Virtual Reality Training in Thyroid Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: G.Gennimatas General Hospital (Other)
Responsible Party: Principal Investigator, Anestis Basios, Principal Investigator, Anestis Basios, G.Gennimatas General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 17010/2910-2024
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Virtual Reality Simulation; Thyroid Surgery
Keywords: Endocrine Surgery; Thyroid Surgery; Virtual Reality; Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): This group will be trained via traditional methods which consists of reading specific chapters of a technical book specialised in Endocrine Surgery (Atlas of Thyroid Surgery- Alexander Shifrin). Also, this group will be provided with videos of the clinic's archive which will support them with specific surgical steps : neck incision up to Continious Neuromonitoring Device placement on Vagus nerve.
  Interventions: Other: Convetional Training
- Virtual Reality Group (Experimental): Participants of this group will be provided with a VR device- MetaQuest3- with an application which will guide them to completion of specific surgical steps from incision up to Continious Neuromonitoring Device placement on Vagus nerve.
  Interventions: Other: Virtual Reality Training in Thyroid Surgery

INTERVENTIONS:
Other: Virtual Reality Training in Thyroid Surgery — Participants will use an application in an Immersive Virtual Reality environment. In this module, the participant will be the chief surgeon and will be guided to accomplise the first steps of thyroidectomy: from neck incision until continious neuromonitoring device placement in vagus nerve.
  Arms: Virtual Reality Group
Other: Convetional Training — This intervation consists of traditional methods of training. Participants will read specific chapters of a technical book specialised in Endocrine Surgery (Atlas of Thyroid Surgery- Alexander Shifrin). Also, they will be provided with videos of the clinic's archive which will support them with specific surgical steps : neck incision up to Continious Neuromonitoring Device placement on Vagus nerve.
  Arms: Control Group

SUMMARY:
Up to this date, there have been no reports on virtual reality (VR) training in thyroid surgery. The purpose of this study is to determine the impact of VR training in residents' education.

Investigators intend to include general surgery residents in the trial, subgrouped in a VR training group and another one with traditional learning, utilizing a technical textbook as a control. For the purpose of this study, a commercial available VR mask will be given for training in the VR group. Randomization will be used to secure balance in the distribution of residents according to their experience. The task which will be examined include surgical steps from neck incision up to the placement of the C-IONM electrode and will be evaluated by a blinded FEBS certified endocrine surgeon in the operating theatre.

Training superiority will be assessed by the outcome measures of Objective Structured Assessment of Technical Skills (OSATS) score, need for the main surgeon to intervene (NTI), verbal answers and time to task completion. Participants will complete questionnaires regarding satisfaction of the whole educational process.

ELIGIBILITY:
Inclusion Criteria:

* Residents of the 2nd Surgical Department of Aristotle University of Thessaloniki
* Residents who have completed their 1st year of training programm.

Exclusion Criteria:

* Disagreement of participants' randomisation
* Prolonged surgical time of completion
* Participant's experience beyond the included limits
* Participants who are completely incapable of using VR devices or have specific helath restrictions of using these
* Patients with complex thyroid disease such as recurrent disease, concominant primary hyperparathyroidism, lymph node disease or metastasis, Graves disease and intrathoracic goiter

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
OSATS Score | From enrollment to the end of assesment of the FEBS certicied surgeon at 1 day
  As the Primary Outcome Measure of the study will be the OSATS(Objective Structured Assessment of Technical Skills) score of participants in each group. Statistical significance of this score between groups will be measured.OSATS is a worlwide tool which measure surgical performance using 7 measurements and scoring system from 7 to 35. Its main advantage is that can measure with a quantitative manner surgical performance.

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Koutelidakis, Professor of Surgery, Study Director — 2nd Surgical Department of Aristotle University of Thessaloniki
Locations (1):
- "Georgios Gennimatas" General Hospital of Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Yes
Any Individual Participant's Data could be shared upon request.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The start date is from enrollment date and end date until study completion

REFERENCES:
- [Background] Ochs V, Saad B, Taha-Mehlitz S, Staubli S, Neumann K, Fischer L, Honaker MD, Lamm S, Rosenberg R, Taha A, Cattin PC. An analysis of virtual reality in abdominal surgery-A scoping review. Int J Med Robot. 2024 Feb;20(1):e2623. doi: 10.1002/rcs.2623. PMID 38375774
- [Background] Rizzetto F, Bernareggi A, Rantas S, Vanzulli A, Vertemati M. Immersive Virtual Reality in surgery and medical education: Diving into the future. Am J Surg. 2020 Oct;220(4):856-857. doi: 10.1016/j.amjsurg.2020.04.033. Epub 2020 Apr 30. No abstract available. PMID 32386709
- [Background] Long AS, Almeida MN, Chong L, Prsic A. Live Virtual Surgery and Virtual Reality in Surgery: Potential Applications in Hand Surgery Education. J Hand Surg Am. 2023 May;48(5):499-505. doi: 10.1016/j.jhsa.2023.01.004. Epub 2023 Feb 9. PMID 36764847
- [Background] Portelli M, Bianco SF, Bezzina T, Abela JE. Virtual reality training compared with apprenticeship training in laparoscopic surgery: a meta-analysis. Ann R Coll Surg Engl. 2020 Nov;102(9):672-684. doi: 10.1308/rcsann.2020.0178. Epub 2020 Aug 21. PMID 32820649
- [Background] Nassar AK, Al-Manaseer F, Knowlton LM, Tuma F. Virtual reality (VR) as a simulation modality for technical skills acquisition. Ann Med Surg (Lond). 2021 Oct 27;71:102945. doi: 10.1016/j.amsu.2021.102945. eCollection 2021 Nov. PMID 34840738
- [Background] Ntakakis G, Plomariti C, Frantzidis C, Antoniou PE, Bamidis PD, Tsoulfas G. Exploring the use of virtual reality in surgical education. World J Transplant. 2023 Feb 18;13(2):36-43. doi: 10.5500/wjt.v13.i2.36. PMID 36908307
- [Background] Mishra R, Narayanan MDK, Umana GE, Montemurro N, Chaurasia B, Deora H. Virtual Reality in Neurosurgery: Beyond Neurosurgical Planning. Int J Environ Res Public Health. 2022 Feb 2;19(3):1719. doi: 10.3390/ijerph19031719. PMID 35162742
- [Background] Falguiere A, LeGruiec C, Herry H, Genest-Beucher S, Dessus JM, Boisrame S. Contribution of virtual reality in oral surgery: A literature review. J Stomatol Oral Maxillofac Surg. 2021 Sep;122(4):405-410. doi: 10.1016/j.jormas.2021.02.004. Epub 2021 Feb 18. PMID 33610770
- [Background] Arjomandi Rad A, Vardanyan R, Thavarajasingam SG, Zubarevich A, Van den Eynde J, Sa MPBO, Zhigalov K, Sardiari Nia P, Ruhparwar A, Weymann A. Extended, virtual and augmented reality in thoracic surgery: a systematic review. Interact Cardiovasc Thorac Surg. 2022 Jan 18;34(2):201-211. doi: 10.1093/icvts/ivab241. PMID 34542639
- [Background] Verhey JT, Haglin JM, Verhey EM, Hartigan DE. Virtual, augmented, and mixed reality applications in orthopedic surgery. Int J Med Robot. 2020 Apr;16(2):e2067. doi: 10.1002/rcs.2067. Epub 2020 Feb 6. PMID 31867864
- [Background] Lohre R, Bois AJ, Athwal GS, Goel DP; Canadian Shoulder and Elbow Society (CSES). Improved Complex Skill Acquisition by Immersive Virtual Reality Training: A Randomized Controlled Trial. J Bone Joint Surg Am. 2020 Mar 18;102(6):e26. doi: 10.2106/JBJS.19.00982. PMID 31972694
- [Background] Lohre R, Bois AJ, Pollock JW, Lapner P, McIlquham K, Athwal GS, Goel DP. Effectiveness of Immersive Virtual Reality on Orthopedic Surgical Skills and Knowledge Acquisition Among Senior Surgical Residents: A Randomized Clinical Trial. JAMA Netw Open. 2020 Dec 1;3(12):e2031217. doi: 10.1001/jamanetworkopen.2020.31217. PMID 33369660
- [Derived] Basios A, Voloudakis N, Atmatzidis S, Velikoudi M, Bellou E, Vamvakidis K, Papaziogas B, Koutelidakis I. The impact of immersive virtual reality training in thyroid surgery: a prospective randomized controlled trial. Updates Surg. 2025 Dec;77(8):2535-2543. doi: 10.1007/s13304-025-02387-8. Epub 2025 Aug 29. PMID 40879873